CLINICAL TRIAL: NCT00478075
Title: A Phase I/II Study of 153 Sm EDTMP (Quadramet™) and PS-341 (Velcade®) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Samarium Sm 153 Lexidronam Pentasodium and Bortezomib in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Angela Dispenzieri, Mayo Clinic Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546736; P30CA015083 (NIH); MC0585 (Other: Mayo Clinic Cancer Center); 1586-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Immunologic Techniques; samarium Sm-153 lexidronam

INTERVENTIONS:
Drug: bortezomib
Other: immunologic technique
Radiation: samarium Sm 153 lexidronam pentasodium

SUMMARY:
RATIONALE: Radioactive drugs, such as samarium Sm 153 lexidronam pentasodium, may carry radiation directly to cancer cells and not harm normal cells. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Bortezomib may also make cancer cells more sensitive to radiation therapy. Giving samarium Sm 153 lexidronam pentasodium together with bortezomib may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of bortezomib when given together with samarium Sm 153 lexidronam pentasodium and to see how well they work in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of bortezomib when given together with samarium Sm 153 lexidronam pentasodium in patients with recurrent or refractory multiple myeloma. (Phase I)
* Determine the safety and tolerability of this regimen in these patients. (Phase II)
* Determine the hematologic response rate in patients treated with this regimen. (Phase II)

Secondary

* Determine the rate of serum immunoglobulin light chain reduction in patients treated with this regimen.
* Assess the in vivo toxicity of this regimen to the progenitor cells by measuring complete blood cell count and micronucleated reticulocyte count in these patients.

OUTLINE: This is a phase I, pilot, open-label, dose-escalation study of bortezomib followed by a phase II study.

* Phase I: Patients receive samarium Sm 153 lexidronam pentasodium IV over 1 minute on day 1 and bortezomib IV over 3-5 seconds on days 2 and 5.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

* Phase II: Patients receive samarium Sm 153 lexidronam pentasodium as in phase I and bortezomib at the MTD determined in phase I .

Patients undergo blood sample collection at baseline and then on days 1-6 for correlative studies. Samples are analyzed for micronucleated reticulocyte count and immunoglobulin free light chain ratio to determine the early effects of treatment.

After completion of study treatment, patients are followed weekly for 7 weeks, monthly for 3 months and then every 3 months for a total of 3 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Relapsed or refractory disease
* Measurable or evaluable disease as defined by at least 1 of the following:

  * Serum monoclonal protein ≥ 1.0 g by protein electrophoresis
  * Monoclonal protein ≥ 200 mg by 24-hour urine electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)
* Previously treated disease

  * No limit to prior therapy provided there is adequate residual organ function
* Must have undergone hematopoietic stem cell collection (for transplant candidates) OR not considered to be a hematopoietic stem cell transplant candidate

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 (ECOG PS of 3 allowed if secondary only to pain)
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* ANC ≥ 1,000/mm^3
* Creatinine ≤ 3 mg/dL
* Calcium ≤ 15 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after completion of study therapy
* No impending long bone fracture
* No other active malignancy except nonmelanoma skin cancer, carcinoma in situ of the cervix, or breast cancer
* No uncontrolled infection
* No known hypersensitivity to any of the components of study drugs
* No other co-morbidity that would preclude study participation

PRIOR CONCURRENT THERAPY:

* Recovered from prior surgery, radiotherapy, or other antineoplastic therapy
* No prior samarium Sm 153 lexidronam pentasodium or strontium chloride Sr 89
* At least 3 weeks since prior myelosuppressive agents
* At least 2 weeks since prior nonmyelosuppressive agents (e.g., thalidomide)
* At least 2 weeks since prior and no concurrent high-dose corticosteroids

  * Chronic steroids (maximum dose of 20 mg/day prednisone or equivalent) allowed for disorders other than myeloma (i.e., adrenal insufficiency or rheumatoid arthritis)
* At least 30 days since prior and no other concurrent investigational therapy
* No concurrent external beam radiotherapy
* No concurrent cytotoxic chemotherapy
* No other concurrent systemic antineoplastic therapy including, but not limited to, any of the following:

  * Immunotherapy
  * Hormonal therapy
  * Monoclonal antibody therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Toxicity (Phase I)
Confirmed clinical response (complete response, very good partial response, partial response, or minimal response) (Phase II)

SECONDARY OUTCOMES:
Immunoglobulin free light chain response
Changes in complete blood cell count and micronucleated reticulocyte count

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, MD, Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Cancer Center, Rochester, Minnesota